CLINICAL TRIAL: NCT01445925
Title: Substrate Modification With Ablation and Antiarrhythmic Drugs in Non-Paroxysmal Atrial Fibrillation
Brief Title: Substrate Ablation and Remodelling in Non-paroxysmal Atrial Fibrillation (AF)
Acronym: SMAAN-PAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dhiraj Gupta, Consultant Cardiologist, Liverpool Heart and Chest Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHCH901
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary vein isolation (Active Comparator): Patients will undergo pulmonary venous isolation plus pharmacological substrate modification
  Interventions: Procedure: Pulmonary vein isolation (PVI); Drug: Pharmacological Substrate modification
- Pulmonary vein isolation + Linear Lesions (Experimental): Patients will undergo pulmonary venous isolation plus both pharmacological and interventional substrate modification
  Interventions: Procedure: Pulmonary vein isolation + linear lesions; Drug: Pharmacological Substrate modification

INTERVENTIONS:
Procedure: Pulmonary vein isolation (PVI) — Using a 4mm irrigated tip radiofrequency ablation catheter a series of lesions >2 mm outside pulmonary vein (PV) ostia will be made to encircle and electrically isolate the pulmonary veins in two ipsilateral pairs (wide area circumferential ablation, WACA). A 20-pole PV mapping catheter will be used to confirm electrical isolation. If the patient is in atrial fibrillation at this stage, sinus rhythm would be restored with electrical cardioversion and PVI would be confirmed in sinus rhythm
  Arms: Pulmonary vein isolation
Procedure: Pulmonary vein isolation + linear lesions — Using a 4mm irrigated tip radiofrequency ablation catheter a series of lesions >2 mm outside PV ostia will be made to encircle and electrically isolate the pulmonary veins in two ipsilateral pairs (wide area circumferential ablation, WACA)34. A 20-pole PV mapping catheter will be used to confirm electrical isolation. Once PVI has been achieved, patients will go onto to receive additional linear ablation lesions. These will include a left atrial roof line, mitral isthmus line, (including ablation inside the coronary sinus if necessary), and ablation on the cavotricuspid isthmus. If the patient is in atrial fibrillation at this stage, the acute end-point would be signal obliteration at the ablated area. Once sinus rhythm is restored with electrical cardioversion, PVI would be confirmed in sinus rhythm and conduction block across the LA roof line, Mitral line and CTI will then be verified with appropriate pacing manoeuvres.
  Arms: Pulmonary vein isolation + Linear Lesions
Drug: Pharmacological Substrate modification — at least 6 weeks therapy with oral amiodarone prior to the ablation procedure and 6 weeks post.

SUMMARY:
The investigators hypothesise that modification of the Atrial Fibrillation (AF) substrate by radiofrequency ablation would improve single procedure success rates for Radio Frequency Ablation (RFA) for Non-paroxysmal AF when compared to that achieved with short-term peri-procedural anti-arrhythmic drug therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing symptoms (European Heart Rhythm Association Class 2 or above) in spite of treatment with rate control medication
* Non-paroxysmal atrial fibrillation, as pre-classified as

  * Persistent AF: AF requiring Electrical/ Chemical cardioversion or that lasting >7 days. These patients may be in AF or in sinus Rhythm at the time of their initial assessment and/ or at the time of their ablation.
  * Continuous Persistent AF: These patients are persistently in AF with or without antiarrhythmic drug therapy, as confirmed on a 24 hour Holter. They may have undergone previous cardioversion(s).
  * Sustained Paroxysmal AF with underlying substrate: Patients with Individual AF episode(s) lasting >12 hours but less than 7 days plus one or more of the following:

    * Age >65 years 21
    * Individual AF episode(s) lasting >24 hours
    * Significant left atrial dilatation of >45 mm on Echo (Parasternal Long Axis view)
    * Obesity (Body Mass Index >30), and/ or history suggestive of sleep apnoea
    * Diabetes Mellitus requiring hypoglycaemic drugs and/or Insulin

Exclusion Criteria:

* Inability or unwillingness to receive oral anticoagulation with warfarin
* Previous Ablation procedure for AF
* Unwillingness or inability to complete the required follow up arrangements
* Presence of long standing persistent AF with continuous AF longer than 12 months. This includes patients in whom sinus rhythm may have been maintained following electrical cardioversion for a period of less than 1 week at a stretch.
* Documented typical atrial flutter
* Prior prosthetic mitral valve replacement or severe structural cardiac abnormality
* Contraindications and/ or prior intolerance to both Amiodarone and Flecainide.
* Reversible cause for atrial fibrillation
* Known hypertrophic or infiltrative cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation/ atrial tachycardia at 6 months following a single procedure. | 12 months
  Defined as >30 sec of AF/ atrial tachycardia identified on ECG or ambulatory ECG monitoring following a 3 month blanking period.

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MD DM MRCP, Principal Investigator — Liverpool Heart and Chest Hospital
Locations (2):
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton and Harefield Hospitals NHS Trust, London

REFERENCES:
- [Derived] Wynn GJ, DAS M, Bonnett LJ, Hall MCS, Snowdon RL, Waktare JEP, Modi S, Todd DM, Gupta D. A novel marker to predict early recurrence after atrial fibrillation ablation: the ablation effectiveness quotient. J Cardiovasc Electrophysiol. 2015 Apr;26(4):397-403. doi: 10.1111/jce.12618. Epub 2015 Feb 25. PMID 25588685